CLINICAL TRIAL: NCT07183566
Title: Ct Volume Measurement of Hepatocellular Carcinoma After Transarterial Chemoembolization (TACE) or Microwave Ablation (MWA)
Brief Title: CT Volume Measurement of Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Saber Hamed Ahmed, Assistant lecturer, Assiut University
Other Study IDs: Ct volume measaurement of HCC
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma (HCC); CT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ct — Ct volume measurement of HCC after TACE or MWA

SUMMARY:
The aim of this study is to evaluate the role of CT volumetric measurement in assessing treatment response of hepatocellular carcinoma (HCC) following trans arterial chemoembolization (TACE) or microwave ablation (MWA)

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the predominant form of primary liver cancer and a major contributor to cancer-related mortality worldwide (1). Conventional curative interventions for HCC encompass liver transplantation, hepatic resection, and thermal ablation. Regrettably, fewer than 30% of patients qualify for surgery upon diagnosis, and many tumor-related characteristics, including size and location, may inhibit the application of thermal ablative methods .

In these cases, locoregional therapies such as transarterial chemoembolization (TACE) and microwave ablation (MWA) play a pivotal role. Both techniques aim to achieve local tumor control and improve patient survival. TACE induces ischemic necrosis through targeted delivery of chemotherapeutic agents combined with arterial embolization, whereas MWA achieves tumor destruction by generating high-frequency electromagnetic waves that produce thermal coagulative necrosis. Accurate assessment of treatment response is essential for guiding clinical decisions and predicting outcomes. Conventional imaging-based response criteria, such as RECIST and mRECIST, primarily focus on changes in lesion diameter. However, these methods may not fully reflect the extent of tumor necrosis or viable residual tissue . In this context, CT-based volumetric measurements have emerged as a more objective and sensitive tool for evaluating therapeutic response after locoregional treatment. Volumetric analysis provides a three-dimensional assessment of tumor burden and may bet ter correlate with treatment efficacy and prognosis compared to traditional linear measurements. Therefore, this study aims to investigate the role of CT volumetric measurement of HCC after TACE or microwave ablation in evaluating treatment response and predicting clinical outcomes .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with a confirmed diagnosis of HCC based on AASLD or EASL criteria.
* Patients deemed unresectable by the multidisciplinary tumor board.
* Patients scheduled for TACE as the primary locoregional therapy.
* Preserved liver function (Child-Pugh class A or B).
* Adequate renal function to permit contrast-enhanced CT.

Exclusion Criteria:

* Patients with extrahepatic metastases or portal vein thrombosis.
* Patients with contraindications to iodinated contrast or TACE.
* Patients with severe comorbid illness that precludes participation.
* Patients refuse to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Assiut University Hospital, Egypt during the period of the study and fulfil the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Ct volume measurent of hepatocellular carcinoma after Transarterial chemoembolization or microwave ablation | Baseline
  At enrollment, all patients will undergo a comprehensive clinical assessment, including full medical history with emphasis on risk factors for hepatocellular carcinoma triphasic CT scan of the liver, which will serve as the reference for tumor volume (by cm3 or cc), number, and distribution prior to TACE or MWA.

IPD SHARING:
Plan to Share IPD: Undecided